CLINICAL TRIAL: NCT01432418
Title: Effectiveness of a Wheelchair Skills Training Program for Power Mobility Users: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lee Kirby, Attending Staff Physician, Department of Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 230378; CDHA-RS/2012-133 (Other: Capital Health Ethics Board)
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Movement Disorders
Keywords: rehabilitation; wheelchairs; safety; disability evaluation; motor skills
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wheelchair training (Experimental)
  Interventions: Other: Wheelchair skills training program
- Control (No Intervention): Standard of care only

INTERVENTIONS:
Other: Wheelchair skills training program — A training program that uses methods based on the rehabilitation, wheelchair, and motor skills literature to teach wheelchair skills.
  Arms: wheelchair training

SUMMARY:
This is a 3-year multi-centre, single-blinded, randomized controlled trial (RCT) to test the hypothesis that wheelchair skills training (using a systematic training program called the Wheelchair Skills Training Program) improves wheelchair skills and safety of 144 powered wheelchair users. A second objective is to assess the effects of age, sex, training centre, and participant experience on outcomes, assessing the retention of benefits and assessing the impact of training on other important outcomes.

ELIGIBILITY:
Inclusion Criteria:

* new or experienced powered wheelchair users
* use or are expected to use powered wheelchairs for at least 4 hrs/week
* have access to a powered wheelchair with a suitable range of controller settings (i.e. able to climb a 5cm level change) for testing and training
* equal or greater than 18 years of age
* able to follow directions in either French or English (whichever is in use at the participating site)
* have the potential to operate their powered wheelchairs independently
* have room for improvement (in the opinion of the potential participant's clinician)
* requires no more than minimal assistance for communication and auditory comprehension (in the opinion of the potential participant's clinician)
* able to follow 2-step commands
* demonstrate the ability to attend training sessions during the intake session
* competent to provide their own informed consent
* able to be comfortably seated in the powered wheelchairs that will be used for the study (if not their own).

Exclusion Criteria:

* use or are expected to use a scooter
* have a rapidly progressive disorder (e.g. amyotrophic lateral sclerosis or terminal cancer)
* have significant visual impairments (legally blind)
* have unstable medical conditions (e.g. angina, seizures)
* have emotional problems (e.g. severe anxiety, depression) that might make participation unsafe or unpleasant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Wheelchair Skills, WST 4.1 questionnaire version | baseline, 1 month , 3 months
  A measure of what the person 'can do' (capacity), 'does do' (performance), and the safety of various wheelchair skills. The Wheelchair Skills Test (WST) version 4.1 in questionnaire format will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD, FRCP, Principal Investigator — Nova Scotia Health Authority
Locations (6):
- Canada (6):
  - GFS Rehabilitation Centre, Vancouver, British Columbia
  - Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia
  - University of Western Ontario, London, Ontario
  - Toronto Rehab, Toronto, Ontario
  - Centre de Réadaptation Lucie-Bruneau, Montreal, Quebec
  - Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale, Québec, Quebec

REFERENCES:
- See also: pubmed Canada study results — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4674291/?tool=nihms